CLINICAL TRIAL: NCT00890370
Title: A Comparison of Five Airway Clearance Techniques in the Treatment of Adults With Cystic Fibrosis
Brief Title: Should Any One Airway Clearance Technique be Recommended for People With Cystic Fibrosis?
Acronym: ACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Dr Jennifer A Pryor, Royal Brompton & Harefield NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1998CF004B
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Airway clearance
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Other): Active cycle of breathing techniques
  Interventions: Procedure: Airway clearance technique
- 2 (Other): Autogenic drainage
  Interventions: Procedure: Airway clearance technique
- 3 (Other): R-C Cornet
  Interventions: Procedure: Airway clearance technique
- 4 (Other): Flutter
  Interventions: Procedure: Airway clearance technique
- 5 (Other): PEP
  Interventions: Procedure: Airway clearance technique

INTERVENTIONS:
Procedure: Airway clearance technique

SUMMARY:
The study was to evaluate the long term effects, over one year, of five airway clearance techniques used by people with cystic fibrosis (active cycle of breathing techniques, autogenic drainage, positive expiratory pressure and oscillating positive expiratory pressure (R-C Cornet and Flutter)). The primary outcome measure was forced expiratory volume in one second (FEV1)and the null hypothesis was that there are no differences among the regimens.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis (genotype or sweat sodium concentration greater than 70 mmol/litre)
* Forced expiratory volume in one second greater than or equal to 25% predicted, on assessment for entry to the study.

Exclusion Criteria:

* Evidence of a current respiratory exacerbation (Thornton et al 2004)
* Current severe haemoptysis
* Past history of pneumothorax
* Awaiting lung / heart-lung transplantation
* Pregnancy
* Recent (within 3 months) acquisition of Burkholderia cepacia

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 1999-07; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | 48 weeks

SECONDARY OUTCOMES:
Quality of life (Short Form-36 and Chronic Respiratory Questionnaire) | 48 weeks
Exercise capacity (Modified shuttle test) | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Pryor, PhD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust